CLINICAL TRIAL: NCT00570349
Title: Safety and Tolerability of Inhaled Nitric Oxide in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INOT 50
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Results first posted 2010-12-01 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2016-05

CONDITIONS: Cystic Fibrosis
Keywords: Inhaled Nitric oxide; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Nitric Oxide; Inhalation; Nitrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose Cohort (Experimental): Subjects in the low dose cohort receive 20 part per million (ppm) of nitric oxide via nasal cannula over a 44 hour period.
  Interventions: Drug: Nitric Oxide for Inhalation
- High-Dose Cohort (Experimental): Subjects in the high dose cohort receive 40 ppm of nitric oxide via nasal cannula over a 44 hour period.
  Interventions: Drug: Nitric Oxide for Inhalation
- Nitrogen (Placebo Comparator): 100% Nitrogen (placebo) will be administer at 20 ppm or 40 ppm via nasal cannula over a 44 hour period.
  Interventions: Drug: Nitrogen

INTERVENTIONS:
Drug: Nitric Oxide for Inhalation — Nitric oxide will be administered at 20 ppm via nasal cannula over a 44 hour period.
  Other Names: INO
  Arms: Low Dose Cohort
Drug: Nitric Oxide for Inhalation — Nitric oxide will be administered at 40 ppm via nasal cannula over a 44 hours period.
  Other Names: INO
  Arms: High-Dose Cohort
Drug: Nitrogen — 100% nitrogen (placebo) will be administered at 20 ppm or 40 ppm via nasal cannula over a 44 hour period.
  Other Names: Nitrogen (N2) Grade 5
  Arms: Nitrogen

SUMMARY:
The primary objective of the trial is to assess the safety and tolerability of inhaled nitric oxide (NO) when administered by nasal cannula over a 44 hour period to clinically stable Cystic Fibrosis (CF) subjects. Toxicity is to be defined as a drop in oxygen saturations, a decline in forced expiratory volume in one second (FEV1), or an increase in methemoglobin.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an autosomal recessive disorder caused by mutations in the gene encoding the cystic fibrosis transmembrane conductance regulator (CFTR) protein. A cycle of chronic, persistent infections with CF-related pathogens and an excessive inflammatory response progressively damages the airways and lung parenchyma, resulting in widespread bronchiectasis and ultimately, respiratory failure. Despite tremendous advances in understanding the CF gene and the CFTR protein, it is not known exactly how mutations in the gene and defects in CFTR lead to persistent airway infection and inflammation.

Inhaled nitric oxide (NO) has potential to be an effective treatment in CF lung disease. Inhaled NO has been studied in other airways diseases characterized by infection and /or inflammation such as COPD and idiopathic pulmonary fibrosis.

NO has been shown to activate CFTR and alternative chloride channels, thereby increasing chloride current in epithelial cells. Therefore, NO treatment may be beneficial in individuals with CF.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* 12 years of age and older
* FEV1 greater than 40% of predicted
* Resting awake oxygen saturation of at least 88%
* Stable pulmonary disease as defined by both clinical impression and having had no recent hospitalizations or changes in antibiotic regimen within 1 month prior to enrollment
* Signed informed consent form

Exclusion Criteria:

* Pulmonary exacerbation resulting in antibiotic treatment (except prophylactic antibiotics) within 1 month of enrollment
* Isolation of B. cepacia from a respiratory tract culture within 6 months
* Severe nasal obstruction at the time of screening
* Receipt of any aerosolized experimental or investigational drugs within 1 month of enrollment
* Pregnancy (a negative pregnancy test must be documented prior to enrollment if applicable)
* Patients who have received treatment with nitric oxide for inhalation within 24 hours prior to study initiation or other investigational medications within 24 hours.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sagel, MD, Principal Investigator — The Children's Hospital
Locations (1):
- The Children's Hospital, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Inhaled Nitric Oxide Low Dose: Low dose group received Inhaled Nitric Oxide at 20 parts per million (ppm) via nasal cannula for 44 hours
- Inhaled Nitric Oxide High Dose: High dose group received Inhaled Nitric Oxide at 40 ppm via nasal cannula for 44 hours.
- Nitrogen: Nitrogen (Placebo) administered at 20 ppm or 40 ppm via nasal cannula over a 44 hour period
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide Low Dose | Inhaled Nitric Oxide High Dose | Nitrogen
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide Low Dose | Inhaled Nitric Oxide High Dose | Nitrogen | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 3 | 13
  Between 18 and 65 years | 1 | 1 | 3 | 5
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.9 (2.14) | 15.6 (2.33) | 17.7 (5.14) | 16.7 (3.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 4 | 4 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Drug, Assessed by Change in Methemoglobin Levels
Description: Methemoglobin level assessments were measured through blood draws - hematology. This test measures the amount of methemoglobin (a type of hemoglobin that is unable to transport oxygen to tissues) in blood. Normal methemoglobin percentage range 1% - 2%.
Time Frame: Baseline and 48 hours
Measure: Mean (Standard Deviation); unit: Percent of Methemoglobin Level
Arm/Group | Inhaled Nitric Oxide Low Dose | Inhaled Nitric Oxide High Dose | Nitrogen
Number analyzed (Participants) | 6 | 6 | 6
Percent of Methemoglobin Level
  Methemoglobin Levels at Baseline | 0.4 (0.14) | 0.5 (0.48) | 0.3 (0.19)
  Methemoglobin Levels at 48 hours | 0.3 (0.14) | 0.1 (0.10) | 0.4 (0.21)

2. Primary Outcome: Change in Oxygen Saturation
Description: Safety and tolerability of drug assessed by decreased oxygen saturation was measured through pulse oximeter, which measure the amount of oxygen in the blood.
  Normal range percentage is 95 - 100%
Time Frame: Baseline and 48 hours
Measure: Mean (Standard Deviation); unit: Percent of oxygen saturation
Arm/Group | Inhaled Nitric Oxide Low Dose | Inhaled Nitric Oxide High Dose | Nitrogen
Number analyzed (Participants) | 6 | 6 | 6
Percent of oxygen saturation
  Oxygen Saturation at Baseline | 95.5 (1.87) | 94.8 (2.14) | 95.5 (2.66)
  Oxygen Saturation at 48 hours | 95.7 (2.16) | 95.8 (3.19) | 97.0 (1.10)

3. Primary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: Decrease in forced expiratory volume in 1 second was measured through spirometer. Spirometer measures the volume of air inspired and expired by the lungs.
Time Frame: Baseline and 48 hours
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Inhaled Nitric Oxide Low Dose | Inhaled Nitric Oxide High Dose | Nitrogen
Number analyzed (Participants) | 6 | 6 | 6
Liters
  Forced Expiratory Volume in 1 second at Baseline | 3.4 (0.66) | 3.1 (1.07) | 3.0 (0.85)
  Forced Expiratory Volume in 1 second at 48 hours | 3.5 (0.66) | 3.1 (1.17) | 3.0 (0.83)

ADVERSE EVENTS:
Arm/Group | Inhaled Nitric Oxide Low Dose | Inhaled Nitric Oxide High Dose | Nitrogen
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide Low Dose (N=6) | Inhaled Nitric Oxide High Dose (N=6) | Nitrogen (N=6)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other